CLINICAL TRIAL: NCT04678505
Title: An Open-Label Trial to Evaluate the Pharmacokinetics of MK-3402 Following Administration of a Single IV Dose to Participants With Mild, Moderate, and Severe Renal Impairment and End-Stage Renal Disease
Brief Title: Study of a Single Intravenous (IV) Dose of MK-3402 in Participants With Impaired Renal Function and in Healthy Controls (MK-3402-004)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3402-004; MK-3402-004 (Other: Merck)
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-04

CONDITIONS: Renal Impairment
Keywords: MK-3402
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Panel A: Mild Renal Impairment (Experimental): Participants with mild renal impairment will receive a single dose of 100 mg MK-3402 via intravenous (IV) infusion on Day 1.
  Interventions: Drug: MK-3402
- Panel B: Moderate Renal Impairment (Experimental): Participants with moderate renal impairment will receive a single dose of 100 mg MK-3402 via IV infusion on Day 1.
  Interventions: Drug: MK-3402
- Panel C: Severe Renal Impairment (Experimental): Participants with severe renal impairment will receive a single dose of 100 mg MK-3402 via IV infusion on Day 1.
  Interventions: Drug: MK-3402
- Panel D: Healthy Participants (Experimental): Healthy matched control participants will receive a single dose of 100 mg MK-3402 via IV infusion on Day 1.
  Interventions: Drug: MK-3402
- Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis (Experimental): Participants with ESRD undergoing HD will receive a single dose of 100 mg MK-3402 via IV infusion after HD on Day 1 of Period 1 and before HD on Day 1 of Period 2. There will be at least a 6-day washout period before dosing in Period 2.
  Interventions: Drug: MK-3402

INTERVENTIONS:
Drug: MK-3402 — MK-3402 administered as a single dose of 100 mg IV infusion on the following dosage days:
  Panels A to D: Day 1 Panel E: Day 1 in Periods 1 and 2

SUMMARY:
The purpose of this study is to compare the plasma and urine pharmacokinetics (PK) of MK-3402 in participants with impaired renal function and healthy control participants, to investigate the extent to which MK-3402 is removed from the plasma by hemodialysis (HD), and evaluate the safety and tolerability of MK-3402 in participants with impaired renal function.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health based on medical history, physical examination, vital signs (VS) measurements, and electrocardiogram (ECG)s performed before randomization.
* Is in good health based on laboratory safety tests obtained at the screening visit and before administration of the initial dose of study drug.
* Has a body mass index (BMI) ≥18 kg/m2 and ≤40 kg/m2. BMI = weight (kg)/height (m)2.
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of study intervention:

  * Refrain from donating sperm
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent or must agree to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause)
* A female participant is eligible to participate if she is a woman of non-childbearing potential.
* Panel A: Has a baseline estimated glomerular filtration rate (eGFR) ≥60 and <90 mL/min/1.73 m2 based on the Modification of Diet in Renal Disease (MDRD) equation.
* Panel B: Has a baseline eGFR ≥30 and <60 mL/min/1.73 m2 based on the MDRD equation.
* Panel C: Has a baseline eGFR ≥15 and <30 mL/min/1.73 m2 based on the MDRD equation.
* Panels A, B and C: Has had no clinically significant change in renal status at least 1 month prior to dosing and is not currently receiving or has not previously been on hemodialysis (HD).
* Panel D: Has an eGFR ≥90 mL/min/1.73 m2 based on the MDRD equation.
* Panel E: Has end stage renal disease (ESRD) and maintained on a stable regimen of at least 3 times per week HD for at least 3 months prior to first dosing.

Exclusion Criteria:

* Panels A, B, C and E: Has a history of any clinically significant concomitant disease or condition (including treatment for such conditions) or diseases whose current condition is considered clinically unstable that, in the opinion of the investigator, could either interfere with the study drug, compromise interpretation of study data, or pose an unacceptable risk to the patient.
* Panel D: Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases. Participants with a remote history of uncomplicated medical events (eg, uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma) may be enrolled in the study at the discretion of the investigator.
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder that would impact study conduct. Participants who have had situational depression may be enrolled in the study at the discretion of the investigator.
* Has a history of cancer (malignancy).

  * Exceptions: (1) Adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or; (2) Other malignancies that have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study, in the opinion of the investigator and with agreement of the Sponsor (eg, malignancies that have been successfully treated ≥10 years prior to the prestudy screening visit).
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or nonprescription drugs or food.
* Is positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Panels A, B, C and E: Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies for the prohibited time period.
* Panel D: Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs or herbal remedies beginning approximately 2 weeks (or 5 half-lives) prior to administration of the initial dose of study drug, throughout the study (including washout intervals between treatment periods), until the poststudy visit. There may be certain medications that are permitted.
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to study drug administration. The window will be derived from the date of the last dose of study medication in the previous study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center ( Site 0001), Orlando, Florida
  - Prism Clinical Research, LLC ( Site 0002), Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male/female participants with mild, moderate, or severe renal impairment (RI), end stage renal disease (ESRD), or healthy matched adults between the ages of 18 and 75 years (inclusive) were recruited at 2 study sites in the United States. However, the study was terminated early due to business reasons prior to enrollment of healthy control participants and participants with severe RI or ESRD, and thus no comparisons could be made.
Groups:
- Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis: Participants with ESRD undergoing hemodialysis (HD) will receive a single dose of 100 mg MK-3402 via IV infusion after HD on Day 1 of Period 1 and before HD on Day 1 of Period 2. There will be at least a 6-day washout period before dosing in Period 2.
Period: Overall Study
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment | Panel C: Severe Renal Impairment | Panel D: Healthy Participants | Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Started | 4 | 5 | 0 | 0 | 0
Completed | 4 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consists of participants in Panels A and B. The study was terminated early due to business reasons prior to enrollment of Panels C, D, and E; thus, no baseline characteristics are presented for healthy control participants and participants with severe RI or ESRD.
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (7.0) | 67.6 (2.6) | 64.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Dosing to Infinity (AUC0-inf) of MK-3402
Description: AUC0-inf is defined as area under the plasma concentration-time curve from dosing to infinity.
Time Frame: Pre-dose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 1
Population: Participants who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model, are included. As the study was terminated early, no participants were enrolled in Panels C, D, or E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µmol/L
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
hr*µmol/L | 71.9 (18.2) | 96.4 (17.5)

2. Primary Outcome: Plasma Concentration at the End of Infusion (Ceoi) of MK-3402
Description: Ceoi is defined as the amount of study drug in plasma following IV infusion administration of study drug. Plasma samples were collected at pre-specified time points and Ceoi was assessed.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
µmol/L | 16.8 (26.0) | 14.3 (31.1)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-3402
Description: Tmax is defined as the time required for a study drug to reach maximum concentration in plasma. Plasma samples were collected at pre-specified time points and Tmax was assessed.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
hours | 0.59 [0.53 to 0.62] | 0.57 [0.55 to 0.75]

4. Primary Outcome: Apparent Plasma Half-life (t½) of MK-3402
Description: t½ is defined as the time required for plasma drug concentration of study drug to decrease by 50% from peak.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
hours | 5.06 (15.2) | 8.12 (9.1)

5. Primary Outcome: Apparent Plasma Clearance (CL) of MK-3402
Description: CL is defined as the time it takes for the study drug to be completely removed from the body's plasma.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
L/hr | 3.13 (18.5) | 2.28 (16.1)

6. Primary Outcome: Volume of Distribution (Vd) of MK-3402
Description: Vd is defined as the distributed volume of study drug in plasma.
Time Frame: Predose and 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
liters | 22.9 (5.3) | 26.6 (20.4)

7. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug
Time Frame: Up to 15 days
Population: All participants who received ≥1 dose of study drug are included. As the study was terminated early, no participants were enrolled in Panels C, D, or E.
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
Participants | 0 | 2

8. Secondary Outcome: Number of Participants Who Discontinued From Study Due to an AE
Description: as for outcome 7
Time Frame: Up to 15 days
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

9. Secondary Outcome: Dialysis Clearance Based on Plasma (CLDplasma) of MK-3402
Description: Plasma dialysis samples were to be collected at pre-specified time points to calculate CLDplasma.
Time Frame: Panel E, Period 2: Pre-dose and 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after the start of infusion
Population: The study was terminated early prior to enrollment of participants on dialysis, and thus no data were collected for this endpoint.
Arm/Group | Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Number analyzed (Participants) | 0

10. Secondary Outcome: Concentration of Dialysate (CD) of MK-3402
Description: Plasma dialysis samples were to be collected at pre-specified time points to calculate CD.
Time Frame: Panel E, Period 2: Pre-dose and 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after the start of infusion
Population: as for outcome 9
Arm/Group | Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Number analyzed (Participants) | 0

11. Secondary Outcome: Amount of Drug Recovered From the Dialysate From Plasma (AED) of MK-3402
Description: Plasma dialysis samples were to be collected at pre-specified time points to calculate AED.
Time Frame: Panel E, Period 2: Pre-dose and 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after the start of infusion
Population: as for outcome 9
Arm/Group | Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Number analyzed (Participants) | 0

12. Secondary Outcome: Percentage of AED (% Dose) of MK-3402
Description: Plasma dialysis samples were to be collected at pre-specified time points to calculate AED (% dose).
Time Frame: Panel E, Period 2: Pre-dose and 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after the start of infusion.
Population: as for outcome 9
Arm/Group | Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Number analyzed (Participants) | 0

13. Secondary Outcome: Hemodialysis Clearance Based on Plasma (CLD Dialysate) of MK-3402
Description: Plasma dialysis samples were to be collected at pre-specified time points to measure CLD dialysate.
Time Frame: Panel E, Period 2: Pre-dose and 1, 1.5, 2, 2.5, 3, 3.5, 4, and 4.5 hours after the start of infusion
Population: as for outcome 9
Arm/Group | Panel E: End-Stage Renal Disease (ESRD) Undergoing Hemodialysis
Number analyzed (Participants) | 0

14. Secondary Outcome: Amount Recovered in Urine From 0 to 24 Hours (Ae0-24) of MK-3402
Description: Ae0-24 is defined as the amount of study drug unchanged in urine after 0-24 hours. Urine samples were collected at pre-specified intervals and Ae0-24 was assessed.
Time Frame: Pre-dose and 0-4, 4-8, 8-12, and 12-24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
mg | 91.8 (32.7) | 61.5 (42.4)

15. Secondary Outcome: Fraction of Dose Recovered in Urine (Fe) of MK-3402
Description: Fe is defined as the fraction of the dose of study drug in urine.
Time Frame: Pre-dose and 0-4, 4-8, 8-12, and 12-24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
percentage | 86.8 (35.1) | 59.7 (41.2)

16. Secondary Outcome: Renal Clearance (CLr) of MK-3402
Description: CLr is defined as the time it takes for the study drug to be completely removed by the kidneys.
Time Frame: Pre-dose and 0-4, 4-8, 8-12, and 12-24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
Number analyzed (Participants) | 4 | 5
L/h | 2.81 (48.6) | 1.52 (36.7)

ADVERSE EVENTS:
Time Frame: Up to 15 days
Description: All participants in Panels A and B who received ≥1 dose of study drug are included. No participants were enrolled into Panels C, D, or E.
Arm/Group | Panel A: Mild Renal Impairment | Panel B: Moderate Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: Mild Renal Impairment (N=4) | Panel B: Moderate Renal Impairment (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)

LIMITATIONS AND CAVEATS:
Due to early study termination, some of the planned endpoints were not able to be completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT04678505/Prot_SAP_000.pdf